CLINICAL TRIAL: NCT02357082
Title: Mayo Clinic Cardiac Implantable Electronic Device (CIED) Magnetic Resonance Imaging (MRI) Registry; Determining the Risks of of MRI in the Presence of Cardiac Implantable Electronic Devices
Brief Title: Mayo Clinic Cardiac Implantable Electronic Device MRI Registry
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert E. Watson, Principal Investigator, Mayo Clinic
Other Study IDs: 14-001925
Record Dates: First submitted 2015-01-20; First posted 2015-02-06 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Magnetic Resonance Imaging
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- MRI Scan: Patients with a previously implanted Cardiac Implantable Electronic Device who are undergoing an MRI Scan for clinically indicated, diagnostic purposes.
  Interventions: Radiation: MRI Scan

INTERVENTIONS:
Radiation: MRI Scan — MRI scan with Specific Absorption Rate (SAR) limit of 1.5 watts per kilogram of body weight
  Other Names: Magnetic Resonance Imaging

SUMMARY:
Registry intends to prospectively collect data regarding the safety of magnetic resonance imaging (MRI) studies in patients with cardiac pacemakers on implantable cardioverter defibrillators.

ELIGIBILITY:
Inclusion Criteria:

* Strong clinical indication for MRI; in the clinical setting where MRI is the diagnostic modality of choice for a specific disease state without acceptable alternative imaging technology
* Male or Female
* 18 years of age or older
* Able to provide informed consent
* Presence of CIED

Exclusion Criteria:

* Presence of metallic objects that represent a contraindication to MR imaging, including: MRI-unsafe intra-orbital or intra-ocular retained metal fragments, and MRI-unsafe intracranial vascular clips and coils, other MRI-unsafe devices
* Morbid obesity (abdominal diameter greater than 60 centimeters) which results in contact wiht the magnet bore.
* Pregnant at time of scanning Pacemaker or Implanted Cardiac Device that is labeled as MRI-Conditional (approved by the Food and Drug Administration for exposure to MRI)
* Pacemaker dependent and either: 1) device implanted before 2005, or 2) advisory pulse generator that may lower outputs in the setting of radiofrequency currents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Mayo Clinic who have a previously implanted CIED and are scheduled for a clinically-indicated MRI will be included in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Cardiac Implantable Electronic Device Lead Impedance at Different Timepoints | Baseline, Visit 1, 3 months, 6 months
Cardiac Implantable Electronic Device Lead Threshold at Different Timepoints | Baseline, Visit 1, 3 months, 6 months
P/R Wave Amplitude at Different Timepoints | Baseline, Visit 1, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Friedman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials